CLINICAL TRIAL: NCT01656109
Title: The Study of Atazavanir/Ritonavir-based HAART in Thai HIV-infected Children
Brief Title: Atazavanir/Ritonavir-based HAART in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); National Health Security Office, Thailand (Other); The Thai Government Pharmaceutical Organization (GPO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 146
Record Dates: First submitted 2012-07-17; First posted 2012-08-02 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: HIV
Keywords: pharmacokinetics; atazanavir/ritonavir; HIV-infected children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PI-experience group (Experimental): Using PI-based HAART for ≥6 months at the screening visit HIV-RNA viral load < 50 copies/ml at the screening visit No history of HIV-RNA ≥ 1,000 copies/ml while using PI-based HAART
  Interventions: Drug: boosted atazanavir (ATV/r)
- PI-naïve group (Experimental): Never been exposed to any PI-containing regimen HIV-RNA viral load ≥ 1,000 copies/ml at the screening visit
  Interventions: Drug: boosted atazanavir (ATV/r)

INTERVENTIONS:
Drug: boosted atazanavir (ATV/r) — ATV/r will be taken orally once daily with food plus standard dose of 2 NRTIs according to Thai National HIV treatment guideline

SUMMARY:
There are no data on efficacy, safety and pharmacokinetics of ATV/r-based HAART in HIV-infected Asian children. Therefore, the investigators aim to evaluate the pharmacokinetics, efficacy and safety of ATV/r-based HAART in Thai HIV-infected children.

DETAILED DESCRIPTION:
Non-nucleoside reverse transcriptase inhibitor (NNRTI)-based HAART have been commonly prescribed as the first-line HAART for HIV-infected children in resource-limited settings. Protease inhibitor (PI)-based HAART are the recommended second-line regimen after failing NNRTI-based HAART. The most commonly used PI in Thailand is lopinavir/ritonavir (LPV/r). However, the metabolic complications of lopinavir/ritonaive (LPV/r) such as hyperlipidemia and lipodyrtrophy are common and a concern for HIV-infected children as it may contribute to the development of cardiovascular disease in the longer term. There are data on efficacy, safety and pharmacokinetics of ATV/r-based HAART in HIV-infected adults but none in children. Furthermore, many studies in both adults and children have shown that different ethnicities can result in different pharmacokinetic response to antiretroviral drugs. As a result of this, this study investigated the efficacy, safety and pharmacokinetics of ATV/r-based HAART in HIV-infected Asian children.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected children
2. Age from 6- 18 years old
3. Body weight ≥ 25 kg at screening visit
4. ARV history, the children can be categorized in one of these 2 groups
5. ALT <200 IU/L at screening visit
6. Total bilirubin < 3 mg/dL at the screening visit
7. Can swallow capsule
8. Written informed consent from caregivers and assent (from children aged 7-17 years who know their HIV status)

Exclusion Criteria:

1. Active opportunistic infection
2. Relevant history or current condition, illness that might interfere with atazanavir/ritonavir absorption, distribution, metabolism or excretion.
3. Use of concomitant medication that may interfere with the pharmacokinetics of ATV/r (i.e. efavirenz, indinavir, proton pump inhibitor, antacids, cisapride, clarithromycin, rifampin etc.)
4. Pregnancy or lactating at screening visit
5. Liver diseases e.g. hepatitis B carrier, chronic hepatitis, cirrhosis
6. Inability to understand the nature and extent of the study and the procedures required.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of atazanavir/ritonavir (ATV/r) | 48 weeks
  Ctrough and Area under the curve (AUC) of atazanavir (ATV) and ritonavir (RTV) will be assessed

SECONDARY OUTCOMES:
CD4 | 48 weeks
  Assess CD percent and count at week 48
plasma viral load (HIV RNA) | 48 weeks
  assess HIV RNA at week 24 and 48
hyperbilirubin | 48 weeks
  evaluate total and direct bilirubin at weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Torsak Bunupuradah, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (3):
- Thailand (3):
  - Department of Pediatrics Faculty of Medicine, Chulalongkorn University, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Division of Infectious Diseases Department of Pediatrics Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok

REFERENCES:
- [Result] Bunupuradah T, Techasaensiri C, Keadpudsa S, Thammajaruk N, Srimuan A, Sahakijpicharn T, Prasitsuebsai W, Ananworanich J, Puthanakit T; HIV-NAT 146 Study Team. Pharmacokinetics of atazanavir/ritonavir among HIV-infected Thai children concomitantly taking tenofovir disoproxil fumarate. Pediatr Infect Dis J. 2014 Dec;33(12):e316-9. doi: 10.1097/INF.0000000000000469. PMID 24983717
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org